CLINICAL TRIAL: NCT07285941
Title: Efficacy and Safety of Distamab Vedotin Combined With Carboplatin for Advanced Ovarian Cancer in the First Line Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, ShaoZhuyan, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCVDTYPEC100
Record Dates: First submitted 2025-09-29; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Cancer; HER2
MeSH Terms: conditions — Ovarian Neoplasms | interventions — RC48 antibody; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): RC48, 2.5 mg/kg, on day 1, every 3 weeks; Carboplatin, AUC 5-6, on day 1, every 3 weeks; q3w, with a maximum of 6 cycles.
  Interventions: Drug: RC48 + Carboplatin

INTERVENTIONS:
Drug: RC48 + Carboplatin — RC48, 2.5 mg/kg, on day 1, every 3 weeks; Carboplatin, AUC 5-6, on day 1, every 3 weeks; q3w, with a maximum of 6 cycles.

SUMMARY:
Ovarian cancer exhibits the highest mortality rate among gynecological malignancies. Currently, the combination of paclitaxel and carboplatin remains the standard first-line chemotherapy regimen for neoadjuvant or postoperative treatment of ovarian cancer. However, conventional paclitaxel, due to the addition of polyoxyethylated castor oil solubilizer, may induce various adverse reactions beyond chemotherapeutic toxicity, such as hypersensitivity, toxic renal injury, neurotoxicity, and cardiovascular toxicity. Therefore, exploring optimized treatment regimens to provide patients with new therapeutic options is imperative.

HER2 is a protein encoded by the ERBB2 gene that regulates cell survival, proliferation, and differentiation. HER2 gene amplification and/or protein overexpression are observed in 18%-35% of mucinous ovarian cancers. A meta-analysis involving over 5,000 ovarian cancer cases revealed that HER2 overexpression correlates with reduced overall survival (OS) and progression-free survival (PFS), suggesting its potential as a biomarker for poor prognosis.

The emergence of novel antibody-drug conjugates (ADCs) has brought new hope for anti-HER2 therapy in ovarian cancer, such as Disitamab Vedotin (RC48). Preliminary results from the PRaG3.0 trial presented at the 2023 ASCO Annual Meeting showed an ORR of 66.7% in six HER2-expressing gynecological cancer patients treated with RC48 combined with radiotherapy and immune checkpoint inhibitors (ICIs). Updated data from the RC48-C018 study demonstrated an ORR of 36.4%, median duration of response (mDoR) of 5.52 months, mPFS of 4.37 months, and 12-month OS rate of 66% in 22 cervical cancer patients. RC48 exhibited promising efficacy and manageable safety in recurrent/metastatic HER2-expressing (IHC 1+/2+/3+) cervical cancer.

Regarding safety, the GOG-158 study reported pronounced hematologic toxicity with carboplatin-paclitaxel in advanced ovarian cancer: grade 3/4 leukopenia (>50%), thrombocytopenia (>30%), and neutropenia (>80%). Conversely, a retrospective study of RC48 combined with platinum ± bevacizumab in HER2-mutated NSCLC patients showed an ORR of 71.4% with no dose reductions or discontinuations due to adverse events. Thus, RC48-platinum combinations may offer a lower-toxicity alternative. Thus the investigators designed this trial to evaluate the efficacy and safety of RC48 combined with carboplatin in HER2-expressing advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Stage II-IV epithelial ovarian cancer, fallopian tube cancer, and primary peritoneal cancer confirmed by histopathological examination;
* Received the first tumor cell debulking surgery before enrollment and achieved R0 or R1 resection;
* HER2 expression: IHC 2+ or 3+;
* Had not received chemotherapy before enrollment;
* ECOG PS ≤ 2;
* Expected survival period ≥ 3 months;
* Adequate organ function. During the screening period, the following criteria should be met (normal values are based on the clinical trial center): Left ventricular ejection fraction ≥ 50%; Hemoglobin ≥ 9 g/dL; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelets ≥ 100 × 109/L; Serum total bilirubin ≤ 1.5 times the upper limit of normal (ULN); When there is no liver metastasis, ALT and AST ≤ 2.5 × ULN, and when there is liver metastasis, ALT and AST ≤ 5 × ULN; Serum creatinine ≤ 1.5 × ULN or calculated creatinine clearance rate (CrCl) ≥ 50 mL/min according to the Cockcroft-Gault formula;
* Non-pregnant women;
* Signed a written informed consent form before the trial.

Exclusion Criteria:

* Within one month prior to the start of treatment, the subject had received other anti-tumor treatments (such as radiotherapy, immunotherapy);
* The subject had central nervous system diseases or brain metastases;
* Had previously experienced grade II or above peripheral neuropathy;
* Had an uncontrolled serious disease that would affect the subject's ability to receive treatment according to the study protocol: such as severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc.;
* Had a history of other malignant tumors within the past 5 years (excluding cured skin basal cell carcinoma and cervical cancer);
* Had known allergies to the study-related drugs or their excipients or was intolerant to them;
* Was participating in other clinical trials at the same time;
* Subjects judged by the researcher to be unsuitable for this study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female
Enrollment: 20 (Estimated)
Dates: Start 2025-01-04 (Actual); Primary Completion 2027-01-04 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
progression free survival | through study completion, an average of 1 year
  The length of time from the start of treatment (or randomisation in a clinical trial) until the disease progresses or the patient dies from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate | up to 12 weeks
  The percentage of subjects who achieved the best response (CR or PR) during the period from the start of the treatment regimen in this study until the onset of disease progression and were excluded from the study, in relation to the total number of subjects in the analyzed dataset.
overall survival | through study completion, an average of 5 year
  It refers to the period from a randomly selected date to the date of death due to any cause.
adverse events | through study completion, an average of 5 year
  Incidence rate of adverse reaction events

CONTACTS AND LOCATIONS:
Locations (1):
- Zhe Jiang Cancer Hospital, Zhejiang, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
To protect participant privacy and confidentiality